CLINICAL TRIAL: NCT01975792
Title: Fetal Thymus Involution as a Predictor of Adverse Neonatal Outcome in Women at High Risk for Preterm Delivery
Brief Title: Fetal Thymus Involution as a Predictor of Adverse Neonatal Outcomes
Acronym: TIPS
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 817255
Record Dates: First submitted 2013-09-04; First posted 2013-11-05 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Women Admitted to Labor and Delivery for the Management of Preterm Labor and/or Preterm Premature Rupture of Membranes (PPROM)
Keywords: PPROM; Pregnant; Preterm; Premature, labor
MeSH Terms: conditions — Preterm Premature Rupture of the Membranes; Premature Birth; Obstetric Labor, Premature

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Preterm Admits: Women who are admitted for preterm labor observation and management

SUMMARY:
The thymus gland is a specialized organ in the chest that plays a central role in the adaptive immune system throughout development until puberty. In response to stress, the fetal thymus gland may shrink, or involute. The investigators propose a prospective cohort study that will enroll pregnant women admitted to labor and delivery for the management of preterm labor and/or preterm premature rupture of membranes from 28-36 weeks gestation. Based on sonographic thymus measurements, the investigators will develop a clinical prediction tool to identify babies who are at increased risk for adverse neonatal outcomes. A reliable non-invasive predictor of adverse neonatal outcome using thymic ultrasound measurements has the potential to affect clinical management, improve outcomes for premature babies, and direct further research efforts.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy between 28-36 weeks gestation
* Active spontaneous preterm labor symptoms (contractions, cervical dilatation and/or PPROM)

Exclusion Criteria:

* Non-singleton pregnancies
* Gestational hypertension/preeclampsia
* Major fetal anomalies
* Known fetal aneuploidy
* Intrauterine Fetal Demise

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant patients with singleton pregnancies admitted to labor and delivery at the Hospital of the University of Pennsylvania between 28-36 weeks gestation for the management of spontaneous preterm labor (defined as uterine contractions and documented cervical change) and/or preterm premature rupture of membranes.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2013-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Respiratory Distress | Date of delivery up to 1 year
  Neonatal respiratory compromise defined as respiratory distress requiring any CPAP (continuous positive airway pressure) and or ventilator therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Nadav Schwartz, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States